CLINICAL TRIAL: NCT00730561
Title: Autologous Hematopoietic Stem Cell Transplantation for the Treatment of Limb Ischemia and Diabetic Neuropathy in Patients With Diabetes Mellitus Type 2:A Randomized Controlled Trial.
Brief Title: Hematopoietic Stem Cell Transplantation for the Treatment of Limb Ischemia and Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Fernando Javier Lavalle Gonzalez, Departamento de Endocrinologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Endo01
Record Dates: First submitted 2008-07-31; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-07

CONDITIONS: Limb Ischemia; Diabetic Neuropathy
Keywords: nerve conduction velocity; hematopoietic stem cell transplantation
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Hematopoietic stem cell transplantation
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Intramuscular application of CD34+ hematopoietic stem cells (with a minimum of 2 million CD34+ cells/kg) into the gastrocnemius muscles after stimulation with subcutaneous filgrastim 600 micrograms/kilogram a day for 4 days
  Arms: 2

SUMMARY:
Several pathophysiological theories have been proposed for the development of diabetic chronic complications. In recent years, the use of stem cells (totipotential, hematopoietic or endothelial lineages) has been reported as an adjunctive modality of treatment for ischemia models in animals and humans. Nevertheless, there are no reports in the use of stem cells for the treatment of human sensorimotor peripheral diabetic neuropathy. We performed this study to evaluate the effect of autologous hematopoietic CD34+ cell transplantation on nerve conduction velocity in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with type 2 diabetes mellitus and ischemia of one or both lower limbs, defined as lack of limb improvement with conventional care (medications, debridements) after a recent amputation or a patient graded III or IV in the Leriche-Fontaine functional classification.

Exclusion Criteria:

* Patients older than 75 years
* Hypercoagulable states
* Cardiac ejection fraction < 30%
* Active vasculopathy in brain, kidneys or heart
* Neoplastic disease
* Active infection
* Diabetic ketoacidosis or hyperosmolar hyperglycemic state
* Gangrene of the extremity requiring immediate surgery.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in nerve conduction velocity | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Lavalle, MD, Principal Investigator — Departamento de Endocrinología del Hospital Universitario "José E. González"
Locations (1):
- Hospital Universitario "José E. González", Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Huang P, Li S, Han M, Xiao Z, Yang R, Han ZC. Autologous transplantation of granulocyte colony-stimulating factor-mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2005 Sep;28(9):2155-60. doi: 10.2337/diacare.28.9.2155. PMID 16123483